CLINICAL TRIAL: NCT06613269
Title: Effect of 68Ga-NY104 and 18F-FDG PET/CT Guided Radiation Therapy Combined with Systemic Treatment in Patients with Clear Cell Renal Cell Carcinoma.
Brief Title: 68Ga-NY104 PET/CT Guided Radiation Therapy in CcRCC.
Acronym: NYCRRT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-413-002
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: clear cell renal cell carcinoma; CAIX; radiation therapy; 68Ga-NY104
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NY104 and FDG guided RT combining systemic therapy (Experimental): In this arm, patients will undergo baseline evaluation using both 68Ga-NY104 and 18F-FGD PET/CT. Metastatic lesions will be identified based on these two PET/CTs and all other imaging modalities available. The radiation field will be planned to cover as much metastasis as possible if not all. Systemic therapy will be delivered at the same time. The patients will be followed up for disease status.
  Interventions: Drug: 68Ga-NY104 PET/CT; Drug: 18F-FDG PET/CT; Radiation: Radiation Therapy; Drug: Systemic therapy

INTERVENTIONS:
Drug: 68Ga-NY104 PET/CT — 68Ga-NY104 PET/CT will be performed at baseline, 6 months, 12 months, and 24 months after radiation therapy if the tumor is under control. If CT or MRI shows any suspicious recurrence or metastasis, 68Ga-NY104 PET/CT can be performed at the decision of the urology oncologist or radiation oncologist.
  The scan begins 1 hour after intravenous injection of 68Ga-NY104.
Drug: 18F-FDG PET/CT — 18F-FDG PET/CT will be performed at baseline and 6 months after radiation therapy. The scan begins 1 hour after intravenous injection of 18F-FDG.
Radiation: Radiation Therapy — Radiation therapy will be delivered to cover as much metastasis as possible if not all. For new lesions after radiation plus systemic therapy, if the new lesions are considered suitable for RT, RT can be delivered again without changing systemic therapy.
Drug: Systemic therapy — Systemic therapy will be delivered to patients to control the tumor. Possible regimen includes targeted therapy alone, immunotherapy alone, and targeted therapy combined with immunotherapy. The treatment regimen will be decided according to the urology oncologist.

SUMMARY:
Radiation therapy (RT) is an effective treatment for patients with advanced-stage clear cell renal cell carcinoma (ccRCC). Current evidence has shown promising outcomes combining radiation therapy and standard systemic therapy in patients with metastatic/recurrent ccRCC. CAIX is a highly sensitive and specific biomarker expressed on ccRCC and in previous studies the investigators have shown excellent diagnostic efficacy of 68Ga-NY104, a CAIX-targeted PET tracer, in patients with metastatic ccRCC. In this study, the investigators aim to investigate the effect of 68Ga-NY104, and 18F-FDG PET/CT guided RT combining standard systemic therapy in patients with metastatic ccRCC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Histologically or cytologically confirmed clear cell renal cell carcinoma
* Eligible for radiation therapy: no more than 10 lesions in total
* Expected survival: over 3 months
* ECOG: 0 or 1
* Sufficient organ function
* Written informed consent

Exclusion Criteria:

* Brain metastasis/carcinomatous meningitis
* Other malignant tumors that are not controlled within 5 years, except for non-metastatic low-risk prostate cancer.
* Pregnant or breastfeeding.
* Active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival 2, PFS2 | the time from the start of RT to 4 years after treatment
  Progression Free Survival 2 (PFS2) was defined as the time from the beginning of treatment to the emergence of new lesions or the progression of original lesions, when the lesions could not be fully covered by radiotherapy, and the drug regimen had to be changed.

SECONDARY OUTCOMES:
Lesion uptake on 68Ga-NY104 PET/CT | From the start of 68Ga-NY104 PET/CT to 1 week after the 68Ga-NY104 PET/CT
Lesion uptake on 18F-FDG PET/CT | From the start of 18F-FDG PET/CT to 1 week after the 18F-FDG PET/CT
Number of positive lesions detected on 68Ga-NY104 PET/CT | From the start of 68Ga-NY104 PET/CT to 1 week after the 68Ga-NY104 PET/CT
Number of positive lesions detected on 18F-FDG PET/CT | From the start of 18F-FDG PET/CT to 1 week after the 18F-FDG PET/CT
Number of lesions detected combining all available imaging modalities | From the start of any imaging modality to 1 week after completion of all imaging modalities
Objective response rate | the time from the start of RT to 4 years after treatment
  The percentage of patients with complete remission or partial remission of tumor after treatment.
Progression free survival 1, PFS1 | the time from the start of RT to 4 years after treatment
  Progression Free Survival 1 (PFS1) was defined as the time from the beginning of treatment to the emergence of new lesions or the progression of original lesions.
Disease control rate | the time from the start of RT to 4 years after treatment
  The percentage of patients with complete remission, partial remission, or stable disease after treatment.
Overall survival | the time from the start of RT to 4 years after treatment
Adverse event | the time from the start of RT to 4 years after treatment
  The adverse event due to PET/CT and treatment will be recorded according to CTCAE 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR